CLINICAL TRIAL: NCT06227611
Title: Evaluation of Different Perimetric Grids to Detect Central Visual Field Defect in Glaucoma Patients with Reduce Ganglion Cell Layer Thickness Measured by Spectral Domain OCT.
Status: Recruiting | Type: Observational
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: GLC04-20
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the study is to evaluate the agreement between three different grids in detecting central visual field defect in early glaucoma patients with reduced ganglion cell layer thickness.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma patients with glaucomatous optic nerve head defect and reduced ganglion cell layer thickness

Exclusion Criteria:

* age<18 years
* unable to read, understand and sign the written informed consent
* unable to perform visual field test
* advanced glaucoma with C/D>0.7
* other causes of optic neuropathies
* retinal or macular diseases
* lens or corneal opacities
* spherical refractive defect >± 6D
* cylindric refractive defect >± 3D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: glaucoma patients referring to glaucoma clinic of IRCCS-Fondazione GB Bietti and University of Rome Tor Vergata.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2025-05-04 (Estimated)

PRIMARY OUTCOMES:
the agreement between 10-2 HFA and 24-2c HFA in detecting central visual field defect | 12 month
  central visual field is defined by the presence of a cluster of three test locations with significantly reduced sensitivity in a hemifield fo the pattern deviation plot.

SECONDARY OUTCOMES:
the agreement between 24-2c HFA and G1 Octopus in detecting central visual field defect | 12 month
  central visual field is defined by the presence of a cluster of three test locations with significantly reduced sensitivity in a hemifield fo the pattern deviation plot.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS-Fondazione GB Bietti, Rome
  - University of Rome Tor Vergata, Rome

IPD SHARING:
Plan to Share IPD: No